CLINICAL TRIAL: NCT07290855
Title: A Phase IV Clinical Study of Evaluating the Safety and Efficacy of Icatibant Injection (Icanticure) in the Treatment of Patients With Bradykinin Induced Angioedema
Brief Title: A Study to Evaluate the Safety and Efficacy of Icatibant in Patients With Bradykinin Induced Angioedema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nang Kuang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKC464-202301
Record Dates: First submitted 2025-03-12; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-03

CONDITIONS: Bradykinin-mediated Angioedema; Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — icatibant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Icatibant Injection (Icanticure®) (Experimental)
  Interventions: Drug: Icatibant Injection (Icanticure®)

INTERVENTIONS:
Drug: Icatibant Injection (Icanticure®) — 30 mg/3 ml injectable prefilled syringe for the treatment of acute attacks of hereditary angioedema (HAE) in children 2 years of age and older.

SUMMARY:
This is a phase IV clinical study. The investigators collect patients with a diagnosis of bradykinin induced angioedema. For a specific study period and prospectively arrange, the eligible patients who has an acute attack of angioedema could be treated by icatibant Injection (Icanticure®).

The drug, icatibant injection has been reimbursed by National Health Insurance Agency, Taiwan (NHI) in the treatment of diagnosed patients with hereditary angioedema. However, the reimbursement is still limited for some patients with atypical conditions. Therefore, Nang Kuang Company initiates a phase IV case collection study and supplies Icanticure® for free during the study period. Patients who still unable to obtain NHI's reimbursed icatibant drug is eligible for the inclusion, enter into the study and can be treated by Icanticure® to meet their clinical urgent needs. The safety and efficacy of Icanticure® are evaluated by the prospective, planed assessments in the enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

1. The male or female patient is ≥20 years old at the time of informed consent.
2. The informed consent form has been read, signed and dated by the patient.
3. At the screening visit, the investigator diagnosed bradykinin-induced angioedema based on at least one of the following:

   * Recurrent attacks of edema and/or poor respond to antihistamines, corticosteroids or epinephrine
   * Recurrent angioedema attacks of abdominal, and/or laryngeal (inclusive of laryngeal and pharyngeal) areas
   * Angioedema without the presence of urticarial rashes
   * Known family history of angioedema
   * Known to have genetic defects related to hereditary angioedema
4. Able to communicate well with the investigator, comply with study questionnaires, and other instruments used for collecting patient-reported outcomes.

Exclusion Criteria:

1. Known with a history of allergy or hypersensitivity to the investigational drug as judged by the investigator at the screening visit.
2. The patient has a diagnosis of angioedema other than bradykinin induced angioedema.
3. The patient has participated in another clinical study within the past 30 days before screening.
4. Presence of liver disease or liver injury as indicated by an abnormal liver function profile such as alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or total bilirubin, if any one of them is out of the reference range.

   The definitions of out of the reference ranges are:
   * Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), or alkaline phosphatase (ALP) > 2.5 times ULN (Upper Limit Normal);
   * Serum total bilirubin >= 1.5 times ULN;
5. Presence of impaired renal function as indicated by abnormal creatinine or blood urea nitrogen values, if any one of them is out of the reference range.

   The definitions of out of the reference ranges are:
   * Creatinine clearance rate (<= 40 mL/min) (estimated by Cockcroft-Gault formula) and serum creatinine >=1.5 times ULN;
   * Blood urea nitrogen value >= 1.5 times ULN
6. Presence of impaired hematological or coagulation functions as indicated by abnormal measure values, if any one of them is out of the reference range.
7. Evidence of symptomatic coronary artery disease based on medical history, in particular, unstable angina pectoris or severe coronary heart disease.
8. Congestive heart failure (NYHA Class 3 and 4).
9. Stroke within the past 6 months.
10. Known pregnancy and/or breast-feeding.
11. In the opinion of the investigator: mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study.
12. In the opinion of the investigator: unlikely to comply with the protocol, for example, uncooperative attitude, inability to return for follow-up visits, or unlikely to complete the study for any reason.
13. In the opinion of the investigator: inability to manage study medication or self-administration of an injection.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
To evaluate the time to complete or near complete resolution from onset of symptoms | Time to complete or near complete resolution of symptoms as reported by the patient, an expected average of 8-10 hours
  The time of onset of acute attack, the time of Icanticure® given, the time of onset of symptom relief, and the time to complete relief of symptoms will be recorded by the patient in minutes. Time to complete relief of symptoms is defined as time from onset of symptoms to complete or near complete resolution as reported by the patient.

SECONDARY OUTCOMES:
Percent Change in VAS pain score: VAS scale ranges from 0-10 with 0 being no any pain and 10 being the highest severity in pain | The time from the onset of acute attack to the time to complete or near complete resolution of symptoms as reported by the patient. The estimated period of time is considered to up to 24 hours.
  The VAS pain scores from 0-10 will be recorded by patients themselves on the following timing, the time of onset of acute attack, the time of Icanticure® given, the time of onset of symptom relief, and the time to complete relief of symptom.
To evaluate volume change of edema from onset of symptoms to complete or near complete resolution. | Volume change will be measured from the onset of acute attack to the time to complete or near complete resolution of symptoms as reported by the patient. The estimated period of time is considered to up to 24 hours
  Volume change of edema will be recorded by patients themselves by using a tape to measure millimeters of the edema part on the following timing, the time of onset of acute attack, the time of Icanticure® given, the time of onset of symptom relief, and the time to complete relief of symptom.
To evaluate the safety and tolerability: the safety profile of Icanticure® will be evaluated by the following parameters. | At least 24 hours post-dose of Icanticure®
  1. Adverse events (AEs) incidence, but the adverse events are not included the pains related to angioedema symptoms which have been evaluated by the VAS pain scores.
  2. Local injection site reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan